CLINICAL TRIAL: NCT03042052
Title: Retrospective Study With Botulinic Toxin in Neurogenic Detrusor Overactivity
Brief Title: Toxin Retrospective Study
Acronym: NDOTOX
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 1637154
Record Dates: First submitted 2017-01-27; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients suffering from NDO managed with Botox: Doses used were 300 units Botox® from January 2001 to January 2011 and 200 units after 2011
  Frequency depended on patient's symptoms
  Duration was an outcome of the study
  Interventions: Drug: detrusor infection of Botulinum toxin

INTERVENTIONS:
Drug: detrusor infection of Botulinum toxin — detrusor injection

SUMMARY:
Aims of this study were to assess the long-term outcomes of detrusor injection of OnabotulinumtoxinA (Botox® injection) associated with clean intermittent-catheterization (CIC) for the treatment of neurogenic detrusor overactivity (NDO) and to identify risk factors for failure.

DETAILED DESCRIPTION:
Neurogenic detrusor overactivity (NDO) remains a major concern for patients with neurological diseases. Fifty to eighty percent of patients with multiple sclerosis (MS) or traumatic spinal cord injury (SCI) and more than 60% of patients with myelomeningocele suffer from urinary incontinence episodes (UI) due to NDO. NDO is characterized by involuntary detrusor contractions during the filling phase, leading to leakage and increase in bladder pressure, which can, precipitate renal failure. Detrusor injection of OnabotulinumtoxinA (Botox®), is licensed worldwide and recommended as a second line therapy for the treatment of urinary incontinence due to NDO after failure of anticholinergic drugs (Grade A).

These recommendations are based on the results of international multicentric, randomized controlled trials.

These studies established not only clinical benefits, with a significant decrease of urinary incontinence episodes, but also urodynamic benefits.

There are very few data about the real prevalence of failure of Botox® in the long term.

Thus, aims of this study were to assess the long-term outcomes of detrusor injections of Botox® associated with clean intermittent-catheterization (CIC) for the treatment of NDO and to identify risk factors for failure .

ELIGIBILITY:
Inclusion Criteria:

* NDO due to MS, SCI or spina-bifida.
* follow-up ≥3 years from the first Botox® injection.
* Performing clean intermittent catheterization

Exclusion Criteria:

* bladder surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from neurogenic detrusor overactivity managed by detrusor injections of Botulinum toxin A and performing clean intermittent catheterization
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
failure ratio | 3 years of follow up
  Survival curves of withdrawals and failures of treatment were calculated with a 95-confidence interval using the Kaplan-Meier method.
Failure ratio | 5 years of follow up
  Survival curves of withdrawals and failures of treatment were calculated with a 95-confidence interval using the Kaplan-Meier method.
Failure ratio | Seven years of follow up
  Survival curves of withdrawals and failures of treatment were calculated with a 95-confidence interval using the Kaplan-Meier method.
withdrawal ratio | 3 years of follow up
  Survival curves of withdrawals and failures of treatment were calculated with a 95-confidence interval using the Kaplan-Meier method.
withdrawal ratio | 5 years of follow up
  Survival curves of withdrawals and failures of treatment were calculated with a 95-confidence interval using the Kaplan-Meier method.
Withdrawal ratio | 7 years of follow up
  Survival curves of withdrawals and failures of treatment were calculated with a 95-confidence interval using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Risk factors for failures based on and clinical, radiological and urodynamic parameters | 3 years
  univariate analysis and multivariate analysis using Cox model
Risk factors for failures based on and clinical, radiological and urodynamic parameters | 5 years
  univariate analysis and multivariate analysis using Cox model
Risk factors for failures based on and clinical, radiological and urodynamic parameters | 7 years
  univariate analysis and multivariate analysis using Cox model

CONTACTS AND LOCATIONS:
Overall Officials: EVEN Alexia, MD, Study Chair — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France

IPD SHARING:
Plan to Share IPD: No